CLINICAL TRIAL: NCT01501877
Title: Smoking Cessation Intervention for Diabetic Patients
Acronym: SSTOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA030532
Record Dates: First submitted 2011-12-21; First posted 2011-12-30 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Smoking; Type 2 Diabetes
Keywords: Smoking; Type 2 Diabetes; Smoking cessation
MeSH Terms: conditions — Smoking; Diabetes Mellitus, Type 2; Smoking Cessation | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Distress Tolerance (Experimental): Acceptance and Commitment Therapy based Distress Tolerance (DT) smoking cessation intervention delivered in 7 2-hour group, 1 50-minute individual, and 2 10-minute phone sessions and 8 weeks of transdermal nicotine patch.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Standard Smoking Cessation (Active Comparator): Standard smoking cessation intervention delivered in 7 2-hour group, 1 50-minute individual, and 2 10-minute phone sessions and 8 weeks of transdermal nicotine patch.
  Interventions: Behavioral: Standard smoking cessation intervention

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — The intervention is based on Acceptance and Commitment Therapy and will be tailored to smokers with Type 2 diabetes.
  Arms: Distress Tolerance
Behavioral: Standard smoking cessation intervention — Standard smoking cessation intervention based on clinical practice guidelines.
  Arms: Standard Smoking Cessation

SUMMARY:
This study is designed to develop and test a smoking cessation intervention for smokers with Type 2 diabetes.

DETAILED DESCRIPTION:
Individuals with Type 2 diabetes smoke at rates similar to those found in the general population, and the health consequences of smoking are particularly severe among smokers with diabetes. In fact, there appears to be a synergistic effect between smoking and diabetes on mortality. However, despite reports that highlight the importance of this work, a paucity of studies have been conducted to develop and test smoking cessation interventions tailored to meet the needs of individuals with diabetes. The small number of extant studies have yielded mixed results. Distress tolerance (DT) focused, acceptance-based interventions have demonstrated efficacy for smoking cessation, and there is increasing support for the conceptual model underlying these interventions among individuals with diabetes. The long-term objective of this research program is to improve smoking cessation treatment for individuals with Type 2 diabetes by developing and establishing the efficacy of a DT smoking cessation intervention tailored to this population. Furthermore, we seek to advance knowledge of the relationships among nicotine withdrawal, negative affect, distress tolerance, and smoking cessation outcomes among individuals with diabetes.

In the present study, we will develop a DT intervention tailored to meet the needs of smokers with Type 2 diabetes. In the first phase of this project, we will develop and pilot the intervention with 18 patients. In the second phase of the project, we will conduct a preliminary, randomized trial with 54 patients to examine the efficacy of the DT intervention relative to a standard smoking cessation treatment (ST) that equates for therapist contact time. Patients in both conditions will receive the transdermal nicotine patch.

We expect that, relative to the ST condition, patients randomized to the DT condition will have increased likelihood of smoking abstinence and increased latency to both smoking lapse and relapse. If the efficacy of this intervention can be established in this trial and in subsequent large scale randomized controlled trials, smokers with diabetes will have improved smoking cessation treatment options. The need for this work is great given the paucity of extant work in this area, the significantly heightened risk of morbidity and mortality from smoking among diabetic patients, the rapidly increasing rate of diabetes in the U.S., and an apparent stabilization of the smoking rate in recent years.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* Type 2 diabetes
* regular smoker for at least 3 years
* smoke an average of more than 10 cigarettes per day
* report motivation to quit smoking of at least 5 out of 10
* speak English

Exclusion Criteria:

* current alcohol abuse or dependence
* current substance abuse or dependence (excluding nicotine)
* psychotic
* form of diabetes other than Type 2
* medical condition that is a contraindication for the transdermal nicotine patch
* using pharmacotherapy for smoking cessation
* using other tobacco products
* unable to provide names and contact information for locators
* no access to a telephone

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Point prevalence abstinence from smoking | 26 weeks from smoking quit date
  We will compare the percentage of participants in each treatment condition who report abstinence from smoking for the 7 days preceding the assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Susan E. Ramsey, Ph.D., Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States